CLINICAL TRIAL: NCT02052362
Title: A Phase I, Open-Label, Single Centre Study Designed to Determine the Absolute Bioavailability of ABT-450 (150 mg) and ABT-267 (25 mg) When Administered as an Oral Co-Formulated Product With Ritonavir (100 mg), ABT 450/r/ABT 267, to Healthy Adult Subjects
Brief Title: Bioavailability of ABT-450 and ABT-267 With Ritonavir
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: M14-229; 2013-003685-14 (EudraCT Number)
Record Dates: First submitted 2014-01-30; First posted 2014-02-03 (Estimated); Last update posted 2014-02-19 (Estimated); Status verified 2014-02

CONDITIONS: Absolute Bioavailability
Keywords: absolute bioavailability; healthy volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 - Regimen A (Experimental): 8 Subjects in Group I - Regimen A: ABT-450/r/ABT-267
  Interventions: Drug: ABT-450/r/ABT-267
- Group 2 - Regimen B (Experimental): 8 Subjects in Group II - Regimen B: ABT-450/r/ABT-267
  Interventions: Drug: ABT-450/r/ABT-267

INTERVENTIONS:
Drug: ABT-450/r/ABT-267 — ABT-450, ABT-267 and ritonavir

SUMMARY:
A study to investigate the fraction of ABT-267 and ABT-450 absorbed by the body when given in combination with each other and Ritonavir(r).

DETAILED DESCRIPTION:
Absolute bioavailability of ABT-267 and ABT-450 in the body when given together

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males or non-pregnant, non-lactating healthy females
2. Body mass index of 18.0 to 30.0 kg/m2
3. Must be willing and able to communicate and participate in the whole study
4. Must provide written informed consent
5. Must agree to use an adequate method of contraception
6. In a condition of general good health, based upon the results of a medical history, physical examination, vital signs, laboratory profile and a 12-lead ECG

Exclusion Criteria:

1. Participation in a clinical research study within the previous 3 months or in an absorption, distribution, metabolism, and excretion (ADME) study within the previous 12 months
2. History of any drug or alcohol abuse in the past 2 years or current smokers and those who have smoked within the last 12 months or a positive cotinine urine test at screening and admission
3. Radiation exposure, including that from the present study, excluding background radiation but including diagnostic x-rays and other medical exposures, exceeding 5 mSv in the last 12 months or 10 mSv in the last 5 years. No occupationally exposed worker, as defined in the Ionising Radiation Regulations 1999, shall participate in the study
4. Positive hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCV Ab) or human immunodeficiency virus (HIV) results
5. Donation or loss of greater than 550 mL of blood (including plasmapheresis) or receipt of a transfusion of any blood product within the previous 8 weeks
6. Subjects who are taking, or have taken, any prescribed or over-the-counter drug or herbal remedies within the 14 days or any drug by injection (including vaccines) within 30 days or within 10 half-lives of the respective medication, whichever is longer, before Investigational Medical Product (IMP) administration

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2014-01; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Absolute bioavailability | Day 1 until 72 hours after single dose of ABT-450/r/ABT-267
  dose normalized AUC(0-inf) for oral dose/dose normalized AUC(0-inf) for IV dose

SECONDARY OUTCOMES:
Safety Labs | Day -1 until 72 hours after single dose of ABT-450/r/ABT-267
  Chemistry, Haematology, Urinalysis
Electrocardiograms (ECGs) | Day-1 until 24 hours after single dose of ABT-450/r/ABT-267
  The measure of any change in 12 lead electrocardiogram from Day-1
Number of participants with adverse events | Screening until 7 days after single dose of ABT-450/r/ABT-267
Physical Exam | Day-1 until 72 hours after single dose ABT-450/r/ABT-267
  To examine any change from Day-1 in the subject's physical presentation (body temperature, blood pressure, pulse)

CONTACTS AND LOCATIONS:
Overall Officials: Armen Asatryan, MD, Study Director — AbbVie
Locations (1):
- Site Reference ID/Investigator# 118615, Nottingham, United Kingdom